CLINICAL TRIAL: NCT05185076
Title: A Prospective, Multicenter, Randomized, Masked, Controlled Pivotal Trial to Assess the Safety and Effectiveness of an Eye-Tracking-Based Treatment for Amblyopia Under Binocular Conditions Versus the Standard of Care, Monocular Deprivation Treatment (Occlusive Patching)
Brief Title: Treatment for Amblyopia Under Binocular Conditions Versus the Standard of Care, Monocular Deprivation Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovaSight (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS-00551
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-12

CONDITIONS: Amblyopia
Keywords: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The EDC and data management will construct a Master Randomization List using a permutated block design stratified by initial visual acuity in the amblyopic eye and age which will specify the order of treatment group assignments. Randomization will be managed directly by the eCRF platform.
Who Masked: Care Provider
Masking Description: Subjects will be seen at follow-up visits. A Masked Examiner must complete distance VA, near VA and stereoacuity testing at these visits. All procedures will be performed with the subject's current spectacle correction. If a subject currently wears spectacles but is not wearing them at the follow-up examination for whatever reason, testing must be performed in trial frames except for Visit 1 and Visit 5 visual acuity must ONLY be performed in current refractive correction glasses (not trial frames).
  Prior to the Masked Examiner entering the room, subjects and parents should be instructed not to discuss their treatment with the Masked Examiner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CureSight eye-tracking-based (Experimental): Device: CureSight Subjects assigned to the binocular treatment group will be prescribed the CureSight treatment to watch for 90 minutes per day, 5 days a week for 16 weeks for the total of 120 hours. Parents of subjects will be instructed that the 90 minutes of daily treatment should be completed in a single 90-minute session, but if this is not possible for whatever reason, the treatment may be divided into two shorter sessions totaling 90 minutes per day
  Interventions: Device: CureSight
- Patching occlusive deprivation (Active Comparator): Device: Patching Subjects assigned to the patching group will wear an adhesive patch over the dominant eye for 2 hours per day, 7 days per week for 16 weeks. Parents of subjects will be instructed that the 2 hours of daily patching should be completed in a single 2-hour session, but if this is not possible for whatever reason, the treatment may be divided into shorter sessions totaling 2 hours.
  Parents will be asked to complete a usage diary by manually recording the patch usage time on daily basis.
  Interventions: Device: CureSight

INTERVENTIONS:
Device: CureSight — watch CureSight treatment for 90 minutes per day, 5 days a week for 16 weeks
  Other Names: Patching ,occlusive deprivation

SUMMARY:
Screening A child is considered for the study after undergoing a standard of care and study specific eye examinations (by a study investigator as part of standard of care) that identifies amblyopia appearing to meet the eligibility criteria. The study will be discussed with the child's parent(s) or guardian(s) (referred to subsequently as parent(s)). Parent(s) who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent / assent must be obtained from a parent and child prior to performing any study-specific procedures that are not part of the child's routine care.

On screening visit, eligibility assessment, medical history,Demographic data, Refraction and Cycloplegia, Demonstration suitability using the CureSight, ATS Diplopia Questionnaire, Symptom Survey Distance VA Testing , Ocular Alignment Testing, Near VA Testing, Stereoacuity Testing-Randot, Stereoacuity Testing- Titmus Fly, Eye movement exams (optional), Contrast sensitivity (optional), Reading rest (optional)

Randomization The EDC and data management will construct a Master Randomization List using a permutated block design stratified by initial visual acuity in the amblyopic eye and age which will specify the order of treatment group assignments. Randomization will be managed directly by the eCRF platform.

All eligible subjects enrolled in the study will be followed for 16 weeks. Subjects will be randomly assigned in a 1:1 allocation to one of the following treatment groups for 16 weeks:

Binocular treatment 90 minutes per day, 5 days per week Patching group: Patching 2 hours per day, 7 days per week. Follow up visits

1-week phone call (4 to 8 days from randomization) to inquire about issues with the CureSight system (if applicable) and to encourage compliance with treatment for all groups (to be completed by site personnel) Visit 2: 4 weeks ± 1 week Visit 3: 8 weeks ± 1 week Visit 4: 12 weeks ± 1 week Visit 5: 16 weeks ± 1 week (primary endpoint) Unmasking of primary outcome results

For each individual subject, clinician's decision regarding:

Treatment or control cessation and follow-up; or, Control (patching) continuation with same modality (more improvement desired); or, Cross-over to a different treatment (avoid missing the optimal window of opportunity in young age)

•Optional Visit 6: 28 weeks ± 1 week (exploratory outcome, including retainment of improvement; and additional exploratory outcomes

DETAILED DESCRIPTION:
Screening A child is considered for the study after undergoing a standard of care and study specific eye examinations (by a study investigator as part of standard of care) that identifies amblyopia appearing to meet the eligibility criteria. The study will be discussed with the child's parent(s) or guardian(s) (referred to subsequently as parent(s)). Parent(s) who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent / assent must be obtained from a parent and child prior to performing any study-specific procedures that are not part of the child's routine care.

On screening visit, eligibility assessment, medical history,Demographic data, Refraction and Cycloplegia, Demonstration suitability using the CureSight, ATS Diplopia Questionnaire, Symptom Survey Distance VA Testing , Ocular Alignment Testing, Near VA Testing, Stereoacuity Testing-Randot, Stereoacuity Testing- Titmus Fly, Eye movement exams (optional), Contrast sensitivity (optional), Reading rest (optional)

Randomization The EDC and data management will construct a Master Randomization List using a permutated block design stratified by initial visual acuity in the amblyopic eye and age which will specify the order of treatment group assignments. Randomization will be managed directly by the eCRF platform.

All eligible subjects enrolled in the study will be followed for 16 weeks. Subjects will be randomly assigned in a 1:1 allocation to one of the following treatment groups for 16 weeks:

Binocular treatment 90 minutes per day, 5 days per week Patching group: Patching 2 hours per day, 7 days per week. Follow up visits

1-week phone call (4 to 8 days from randomization) to inquire about issues with the CureSight system (if applicable) and to encourage compliance with treatment for all groups (to be completed by site personnel) Visit 2: 4 weeks ± 1 week Visit 3: 8 weeks ± 1 week Visit 4: 12 weeks ± 1 week Visit 5: 16 weeks ± 1 week (primary endpoint) Unmasking of primary outcome results

For each individual subject, clinician's decision regarding:

Treatment or control cessation and follow-up; or, Control (patching) continuation with same modality (more improvement desired); or, Cross-over to a different treatment (avoid missing the optimal window of opportunity in young age)

•Optional Visit 6: 28 weeks ± 1 week (exploratory outcome, including retainment of improvement; and additional exploratory outcomes)

The call center will be comprised of NovaSight personnel, protected by a firewall. For the patching group subjects, the call center personnel will contact all subjects' guardians at 1 week (3 to 7 days) to encourage initial compliance with treatment.

For the CureSight treatment group, the call center will contact the subjects' guardians in order to:

Assist first time setup at home over the phone Provide technical support by phone in case of system malfunction or any other query or problem appearing during treatment Respond to compliance notifications of the software and contact the subject's guardians when needed in order to encourage compliance Answer any questions that arise by the subjects or guardians. Permission for such contacts will be included in the Informed Consent Form.

The call center personal will be exposed to the following details, contact information, email and phone number.

ELIGIBILITY:
The following criteria must be met for a child to be enrolled in the study:

1. Age 4 to <9 years male and female
2. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated)

   1. Criteria for strabismic amblyopia: At least one of the following must be met:

      * Presence of a heterotropia on examination at distance or near fixation (with or without optical correction, must be no more than 5 PD by SPCT at near fixation
      * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)
   2. Criteria for anisometropia: At least one of the following criteria must be met:

      * ≥1.00 D difference between eyes in spherical equivalent
      * ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes
   3. Criteria for combined-mechanism amblyopia: Both of the following criteria must be met:

      * Criteria for strabismus are met (see above)
      * ≥1.00 D difference between eyes in spherical equivalent OR ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes

   Amblyopia associated with anisometropia, strabismus or both meeting at least one of the following conditions:
   * Newly diagnosed amblyopia (i.e. no prior treatment)
   * If there had been prior amblyopia treatment, it must have been discontinued with no treatment administered for Non- a minimum of 8 weeks prior to the Screening Visit
3. Must have refractive error correction (based on a cycloplegic refraction completed within the last 7 months) if any of the following are true:

   * Hypermetropia of 2.50 D or more by spherical equivalent (SE)
   * Myopia of amblyopic eye of 0.50D or more SE
   * Astigmatism of 1.00D or more
   * Anisometropia of more than 0.50D SE NOTE: Subjects with cycloplegic refractive errors that do not fall within the requirements above for spectacle correction may be given spectacles at investigator's discretion, but must follow the study-specified prescribing guidelines, as detailed below.

     c. Spectacle prescribing instructions referenced to the cycloplegic refraction completed within the last 7 months:
   * SE must be within 0.50D of fully correcting the anisometropia.
   * SE must not be under corrected by more than 1.50D SE, and reduction in plus sphere must be symmetric in the two eyes.
   * Cylinder power in both eyes must be within 0.50D of fully correcting the astigmatism.
   * Axis must be within +/- 10 degrees if cylinder power is ≤1.00D, and within +/- 5 degrees if cylinder power is >1.00D.
   * Myopia must not be under corrected by more than 0.25D or over corrected by more than 0.50D SE, and any change must be symmetrical in the two eyes.

     d. Spectacle correction meeting the above criteria must be worn:
   * For at least 16 weeks OR until distance VA stability is documented (defined as <0.1 logMAR change by the same testing method measured on 2 consecutive exams at least 8 weeks apart).
   * For determining VA stability (non-improvement):

     * The first of two measurements may be made 1) in current spectacles, or 2) in trial frames with or without cycloplegia or 3) without correction (if new correction is prescribed),
     * The second measurement must be made without cycloplegia in the correct spectacles that have been worn for at least 8 weeks.
     * Note: since this determination is a pre-study procedure, the method of measuring VA is not mandated.
4. VA, measured in each eye without cycloplegia in current spectacle correction (if applicable) within 7 days prior to randomization using the Lea symbol per ATS VA protocol for children < 7 years and the E-ETDRS VA protocol for children ≥ 7 years on a study-approved device displaying single surrounded optotypes, as follows:

   1. Visual acuity in the amblyopic eye 20/32 to 20/100 inclusive
   2. Best-corrected dominant-eye VA meeting the following criteria:

      * If age 4, 20/40 or better by Lea symbol per ATS
      * If age 5 and older, 20/32 or better by ATS-HOTV using LEA symbols for age <7 and Lea numbers for > 7 years
   3. Interocular difference ≥ 2 logMAR lines (Lea symbol per ATS)
5. Heterotropia with a near deviation of <5∆ (measured by SPCT) in habitual correction (Angles of ocular deviation >4∆ are not allowed because large magnitudes of the deviation would compromise successful alignment of the dichoptic stimuli.)
6. Passing a dedicated 10 min in-clinic performance ability test to assure suitable eye tracking performance (validity of eye tracking data >90% and successful calibration process).
7. Subjects and families eligible for clinic visits over duration of study.
8. Subject in general good health and able, as per investigator decision, to comply with study visits and protocol procedures and wear refractive correction and has access to wireless internet at home which is able to support the CureSight treatment (loaned by sponsor).
9. Signed and dated informed consent form.
10. Parent and participant understand and are willing to comply with study procedures and will be available for the duration of the study.

Exclusion Criteria

A subject is excluded for any of the following reasons:

1. Myopia greater than -6.00 D. spherical equivalent in either eye.
2. Known skin reactions to patch or bandage adhesives.
3. Any other condition which could be a potential cause for reduced BCVA according to the investigator.
4. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Subjects with mild speech delay or reading and/or learning disabilities are not excluded.
5. History of low adherence with amblyopia treatment as assessed informally by the investigator.
6. Subjects that do not wear their spectacles. (as assessed by investigator)
7. History of light-induced seizures.
8. Wearing RGP contact lenses.
9. Any reported anatomic ocular anomaly (e.g., small lens opacity, myelinated nerve fiber layer).
10. Previous intraocular or refractive surgery.
11. Any condition that prevents the subject from completing a continues 45-90 min. of treatment per day while seating in front of a near screen. Such as children who don't like or cannot watch TV/movies for more than 60 min every day according to the parent's report.
12. Heterophoria with a total near deviation of ≥10Δ (measured by PACT).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | 16 weeks
  mean change in amblyopic eye distance BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Spierer, MD, Principal Investigator — Tel Aviv University
Locations (2):
- Israel (2):
  - Rambam medical center, Haifa
  - Haim Sheba medical center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wygnanski-Jaffe T, Moshkovitz A, Kushner BJ, Belkin M, Yehezkel O; CureSight Pivotal Trial Group. Binocular Home Treatment for Amblyopia: Gains Stable for One Year. Am J Ophthalmol. 2024 Jun;262:199-205. doi: 10.1016/j.ajo.2024.02.004. Epub 2024 Feb 14. PMID 38360334